CLINICAL TRIAL: NCT03607357
Title: The Effect of Post-extubation High Flow Nasal Oxygen in Patients With Acute Left Heart Failure: a Clinical Multi-center Study
Brief Title: High Flow Nasal Oxygen and Acute Left Heart Failure
Acronym: HFNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Jiangbei People's Hospital (Other)
Collaborators: Jiangsu Provincial People's Hospital (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); NanJing PLA 81 Hospital (Other); Nanjing Chest Hospital (Unknown); Mingji Hospital (Other); Meishan Traditional Chinese Medicine Hospital (Other); Nanjing LuHe People's Hospital (Unknown); Nanjing Pukou Center Hospital (Other); Thank Inn Chain Hotel Jiangsu Nanjing Lishui People's Hospital (Other); Nanjing Gaochun People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018020
Record Dates: First submitted 2018-07-02; First posted 2018-07-31 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure; Noninvasive Ventilation; Oxygen Therapy
Keywords: High Flow Nasal Oxygen; Non-invasive Ventilation; Acute Left Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNO group/Group A (Experimental): The patients should receive the treatment of high flow nasal oxygen immediately after extubation.
  Interventions: Device: High Flow Nasal Oxygen
- NIV group/Group B (Placebo Comparator): The patients should receive the treatment of non-invasive Ventilation immediately after extubation.
  Interventions: Device: Non-invasive Ventilation

INTERVENTIONS:
Device: High Flow Nasal Oxygen — The initial flow speed is set at 30L/min and increases at 5L/min in titrated type until the patient feels uncomfortable. The temperature is set at 37℃. The fraction of inspiration O2 is set in accordance with specific condition of patient to insure oxygen saturation more than 95%.
  Arms: HFNO group/Group A
Device: Non-invasive Ventilation — The values of initial pressure are set at a lower level (inspiratory pressure: 6-8cmH2O, expiratory pressure: 4cmH2O) and adjusted to a suitable level in 10-20min. The fraction of inspiration O2 is set in accordance with specific condition of patient to insure oxygen saturation more than 95%.
  Arms: NIV group/Group B

SUMMARY:
Acute left heart failure (ALHF) is a sudden attack or deterioration of abnormal left heart function, which may impair myocardial contractility and increase cardiac loading, further result in decreased cardiac output, abrupt elevation of pulmonary and systemic circulation pressure, consequently trigger in acute pulmonary congestion, acute pulmonary edema and cardiac shock .

Hypoxia and severe dyspnea may pose fatal threats for the patients suffered from ALHF should be alleviated as soon as possible, and thus oxygen therapy and ventilation support are regarded as important therapeutic measures for these patients. According to 2017 Chinese College of Emergency Physicians(CCEP) acute heart failure clinical guideline, invasive ventilation should be recommended to those patients whose symptoms still get worsening despite timely treatments.

Intubation may increase the risks of infection and multiple organ failure, so timely extubation contributes to reduce the duration of mechanical ventilation and the rate of complications. But if extubation failure occurs, the patient often requires re-intubation that may induce the outset of complications, extend the length of stay and increase mortality.

Heart failure proves to be high risk factor for extubation failure on the basis of previous studies. It is recommended to apply sequential non-invasive ventilation (NIV) if the patient receiving invasive ventilation for more than 24 hours and having high risk for extubation failure on the basis of 2017 American Thoracic Society(ATS) clinical guideline. It is worthy to note that NIV has many shortcomings, for example, it may induce dry oropharyngeal cavity, skin injury caused by mask oppression, gaseous distention, vomiting, respiratory aspiration, air leak, drying sputum, difficulty in coughing up phlegm and claustrophobia.

As an emerging technology, high flow nasal oxygen (HFNO) has many advantages in airway humidification, tolerance and compliance which also can effectively improve pulmonary oxygenation function of patients with respiratory failure. Which therapeutic measure should be recommended for the patients with ALHF after extubation, NIV or HFNO? It is still unclear according to the latest management guidelines. So one perspective study will be launch to compare the difference between HFNO-group patients with NIV-group patients in re-intubation rate within 48 hours, oxygenation index, length of ICU stay, total hospital stay, mortality and compliance for evidence-based medicine.

DETAILED DESCRIPTION:
1. The anticipated number of patient subjects will reach 120 in the study. The patient's condition should be informed to his/her next of kin and then agree to signs the informed consent.
2. When passing spontaneous breathing trials and removing tracheal tube, the patients should be divided into two groups by random digital table.
3. Group A/HFNO group: the patients should receive the treatment of high flow nasal oxygen immediately after extubation. The initial flow speed was set at 30L/min and increased at 5L/min in titrated type until the patient feels uncomfortable. The temperature was set at 37℃. The fraction of inspiration O2 was set in accordance with specific condition of patient to insure oxygen saturation more than 95%.

   Group B/NIV group: the patients should receive the treatment of non-invasive ventilation immediately after extubation. The initial pressure are set at a lower level (inspiratory pressure: 6-8cmH2O, expiratory pressure: 4cmH2O) and adjusted to a suitable level in 10-20min. The fraction of inspiration O2 was set in accordance with specific condition of patient to insure oxygen saturation more than 95%.
4. The criteria of successful extubation: the patient doesn't require re-intubation within 48 hours after extubation.

   The criteria of extubation failure: the patient needs re-intubation and ventilation support within 48 hours after extubation.
5. (1) Investigators should keep a record of these patient's general condition, for instance, age, sex, diagnosis, Apache II score, treatment, etc.(2) Investigators should routinely detect clinical manifestation, ventilation parameters and physiological indices of the recruited patients. Elementary monitoring indicators consist of vital signs, oxygen saturation, ECG, tidal volume, breathing rate, inspiratory pressure, expiratory pressure and blood gas analysis. Blood gas analysis should be evaluated on an average of 12 hours, within the range of 48 hours after extubation.(3) Clinical prognosis of these patients should be recorded, including the rate of weaning failure, re-intubation rate, time for re-intubation, causes of re-intubation, duration of HFNO/HIV, length of ICU stay, hospitalization time and number of death.（4） The data of adverse effect derived from devices applied in the study should be recorded. HFNO group: dry nasal cavity, dry oropharyngeal cavity, dysphagia.HIV group: dry oropharyngeal cavity, skin injury caused by mask oppression, gaseous distention, vomiting, respiratory aspiration, air leak, drying sputum, difficulty in coughing up phlegm and claustrophobia.

ELIGIBILITY:
Inclusion Criteria:

* (1) Clinical diagnosis of acute left heart failure
* (2) The patient receives invasive ventilation for more than 24 hours
* (3) Must pass spontaneous breathing trials
* (4) Patient's next of kin agrees to sign the informed consent.

Exclusion Criteria:

* (1) Chronic Obstructive Pulmonary Disease (COPD)
* (2) Disturbance of consciousness
* (3)Bulbar paralysis, dysphagia
* (4) Facial deformity
* (5) Terminal tumor
* (6) Neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
re-intubation rate within 48 hours | 48 hours after extubation.

SECONDARY OUTCOMES:
Mortality | 28 days after joining the study.
Hospitalization time | From date of randomization to the day when the patient discharges from any cause, assessed up to three months
The length of ICU stay | From date of randomization to the day when the patient leaves ICU ward, assessed up to three months
blood gas analysis | on an average of 12 hours, within the range of 48 hours after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Zhenglong Ye, bachelor, Study Director — Nanjing Jiangbei People's Hospital
Locations (1):
- Nanjing Jiangbei People's Hospital, Nanjing, Jiangsu, China